CLINICAL TRIAL: NCT00999700
Title: Induction Chemotherapy Followed by Cetuximab Plus Definitive Radiotherapy Versus Radiation Plus Cisplatin
Acronym: INTERCEPTOR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Principal Investigator, MARCO MERLANO, MD, Gruppo Oncologico del Nord-Ovest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT NUMBER 2009-013402-14
Record Dates: First submitted 2009-10-16; First posted 2009-10-22 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Locally advanced HNSCC; Chemo-radiation; Induction chemotherapy; Stage III/IV; Unresectable disease
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy; Cetuximab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A (Experimental): Induction chemotherapy: TCF (Vermorken, N Eng J Med 2007) Definitive treatment: RT + C-mab (Bonner, N Eng J Med 2006)
  Interventions: Drug: docetaxel - cisplatin - 5-fluorouracil; Radiation: radiotherapy; Drug: cetuximab
- ARM B (Active Comparator): RT + Cddp (RTOG, Adelstein, J Clin Oncol 2003)
  Interventions: Drug: cisplatin; Radiation: radiotherapy

INTERVENTIONS:
Drug: docetaxel - cisplatin - 5-fluorouracil — docetaxel 75 mg/sqm day1 cisplatin 75 mg/sqm day1 5-fluorouracil 750 mg/sqm/d c.i. day1 to day4 q21
  Arms: ARM A
Radiation: radiotherapy — Conformal radiotherapy or IMRT should be employed.
  Standard radiotherapy:
  Minimum radiation dose 70 Gy. Additional boost up to 10 Gy if clinically indicated.
  Arms: ARM A
Drug: cetuximab — 400 mg/sqm at the 1st infusion - before starting RT 250 mg/sqm weekly - concurrent with RT up to the last week of treatment
  Arms: ARM A
Drug: cisplatin — Cisplatin, 100 mg/sqm every 3 weeks, three times, concurrent with RT, starting from day 1 of treatment.
  Arms: ARM B
Radiation: radiotherapy — Conformal radiotherapy or IMRT should be employed.
  Standard radiotherapy:
  Minimum radiation dose 70 Gy. Additional boost up to 10 Gy if clinically indicated.
  Arms: ARM B

SUMMARY:
A phase III trial of induction chemotherapy followed by definitive radiotherapy plus Cetuximab versus chemoradiation in unresectable, locally advanced, squamous cell carcinoma of the head and neck (HNC).

DETAILED DESCRIPTION:
The objective of this trial is to determine whether Cetuximab and radiation preceded by an induction chemotherapy, may be superior to an established chemoradiation program for HNC (RTOG regimen, Adelstein DJ J.Clin.Oncol. 2003;21:92-98).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Histologically or cytologically confirmed diagnosis of HNSCC
* Stage III/IV, not suitable for surgery (definitive cure rate improbable, technically unresectable or medical contraindication for surgery)
* At least one uni-dimensional measurable lesion either by CT scan or MRI
* Signed written informed consents prior to beginning protocol

Specific procedures:

* Tumor tissue available for immunohistochemical staining of EGFR expression and HPV
* Life expectancy of > 3 months at study entry
* ECOG Performance Status of <2 at study entry.
* Effective contraception if risk of conception exists.
* Neutrophils > 2.0/mm³, platelet count > 100,000/mm³, and hemoglobin > 10 g/dl
* Normal liver function
* Serum creatinine > 1.25 x ULN and/or creatinine clearance > 60 ml/min

Exclusion Criteria:

* Prior systemic chemotherapy and/or radiotherapy
* Known peripheral neuropathy > grade 2 NCI-CTC version 3.0
* Known chronic heart failure
* Prior surgery, excluding prior diagnostic biopsy
* Known drug abuse
* Active uncontrolled infection
* Other concomitant anticancer therapy
* Distant metastasis
* Concurrent chronic systemic immune therapy, chemotherapy for disease other than cancer, or hormone therapy not indicated in the study protocol
* Clinically relevant coronary artery disease or history of a myocardial infarction within the last 12 months before study entry
* Medical or psychological condition that would not permit the patient to complete the trial or sign informed consent
* Nasopharyngeal carcinoma WHO type II or III
* Known allergic reaction against any of the components of the treatment
* Pregnancy (absence confirmed by beta-HCG test) or lactation period
* Any prior or on-going investigational medication
* Previous or current malignancy except basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2009-09; Primary Completion 2016-12-31 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years

SECONDARY OUTCOMES:
Incidence of acute and late toxicities in the two arms | 5 years
Progression free survival | 5 years
Locoregional control | 5 years
Response rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: MARCO MERLANO, MD, Principal Investigator — ASCO, ESMO, AIOM, G.O.N.O.
Locations (21):
- Italy (21):
  - Ospedale S. Giacomo, Novi Ligure (al), Italy
  - Irccs Centro Di Riferimento Oncologico Di Basilicata (Crob), Rionero in Vulture (pz), Italy
  - Ospedale Civile Ss. Antonio E Biagio, Alessandria
  - Ausl Della Valle D' Aosta, Aosta
  - Policlinico S. Orsola-Malpighi, Bologna
  - Asl 8 - Ospedale Businco, Cagliari
  - A.S.O. S. Croce E Carle, Cuneo
  - Irccs - Aou S. Martino - Oncology, Genoa
  - Irccs - Aou San Martino - Radiotherapy, Genoa
  - Asl 3 Genovese, Genova
  - E.O. Ospedali Galliera, Genova
  - Azienda Ospedaliera Villa Scassi - Asl3, Italy
  - Istituto Nazionale Dei Tumori, Milan
  - Azienda Ospedaliero Universitaria Di Modena, Modena
  - Azienda Ospedaliero-Universitaria Di Parma, Parma
  - Azienda Ospedaliera Ospedali Riuniti Di Fano, Pesaro
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale S. Filippo Neri, Roma
  - Ospedale S. Paolo, Savona
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino Torino (to), Turin
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino, Turin

REFERENCES:
- [Result] - J.P. Pignon et al. Lancet 2000
- [Result] - A. Forastiere et al., New Engl J Med 2001
- [Result] - Adelstein DJ J.Clin.Oncol. 2003
- [Result] - Henke, New England 2004
- [Result] - J.A. Bonner et al., New Engl J Med 2006
- [Result] Merlano M. Alternating chemotherapy and radiotherapy in locally advanced head and neck cancer: an alternative? Oncologist. 2006 Feb;11(2):146-51. doi: 10.1634/theoncologist.11-2-146. PMID 16476835
- [Result] - Posner M et al, New Engl J Med 2007
- [Result] - Vermorken J et al, New Engl J Med 2007
- [Result] - Lo Nigro, Journal of Cancer Research Clinical Oncology 2009
- [Result] Merlano M, Marchetti G. Radiochemotherapy in head and neck cancer. Cancer Treat Rev. 2003 Aug;29(4):291-6. doi: 10.1016/s0305-7372(03)00022-7. PMID 12927569
- See also: click on "trials" for more informations — http://www.reteoncologica.it/